CLINICAL TRIAL: NCT00851994
Title: Urine Proteome of Patients Undergoing Surgery
Brief Title: Urine Proteome of Patients Having Surgery
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201103022
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Surgery
Keywords: Patients having surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting urine and blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients having surgery

SUMMARY:
The investigators are measuring novel proteins in the urine of patients having surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Undergoing surgery

Exclusion Criteria:

* No formal exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having surgery.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2008-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in urine proteins after surgery. | Pre-op, intraoperative, post operatively (1-6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Morrissey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Hu R, Gupta R, Wang Z, Wang C, Sun H, Singamaneni S, Kharasch ED, Morrissey JJ. Bioplasmonic paper-based assay for perilipin-2 non-invasively detects renal cancer. Kidney Int. 2019 Dec;96(6):1417-1421. doi: 10.1016/j.kint.2019.08.020. Epub 2019 Sep 3. PMID 31668633
- [Derived] Morrissey JJ, Mobley J, Figenshau RS, Vetter J, Bhayani S, Kharasch ED. Urine aquaporin 1 and perilipin 2 differentiate renal carcinomas from other imaged renal masses and bladder and prostate cancer. Mayo Clin Proc. 2015 Jan;90(1):35-42. doi: 10.1016/j.mayocp.2014.10.005. PMID 25572193
- [Derived] Morrissey JJ, Kharasch ED. The specificity of urinary aquaporin 1 and perilipin 2 to screen for renal cell carcinoma. J Urol. 2013 May;189(5):1913-20. doi: 10.1016/j.juro.2012.11.034. Epub 2012 Nov 12. PMID 23154208
- [Derived] Morrissey JJ, London AN, Lambert MC, Kharasch ED. Sensitivity and specificity of urinary neutrophil gelatinase-associated lipocalin and kidney injury molecule-1 for the diagnosis of renal cell carcinoma. Am J Nephrol. 2011;34(5):391-8. doi: 10.1159/000330851. Epub 2011 Sep 7. PMID 21912102
- [Derived] Morrissey JJ, London AN, Luo J, Kharasch ED. Urinary biomarkers for the early diagnosis of kidney cancer. Mayo Clin Proc. 2010 May;85(5):413-21. doi: 10.4065/mcp.2009.0709. Epub 2010 Apr 7. PMID 20375178